CLINICAL TRIAL: NCT04641728
Title: A Phase 2 Study of Pembrolizumab in Combination With Olaparib in Patients With Recurrent or Metastatic Cervical Cancer Who Had Disease Progression During or After Platinum-based Chemotherapy
Brief Title: Pembrolizumab Plus Olaparib in Patients With Recurrent Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saitama Medical University International Medical Center (Other)
Collaborators: Tokyo University (Other); National Cancer Center, Japan (Other Government); Cancer Institute Hospital, Japan (Other); Aichi Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOTIC-025
Record Dates: First submitted 2020-11-02; First posted 2020-11-24 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-07

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; pembrolizumab; olaparib
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — pembrolizumab; olaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- pembrolizumab plus olaparib (Experimental): Until RECIST-based confirmation of progressive disease (PD), death, manifestation of intolerable toxicity, or participant withdrawal from the study, study participants will continue intravenous infusion of pembrolizumab 200 mg every three weeks (Q3W) in combination with oral olaparib 300 mg twice daily (BID) (combination therapy)
  Interventions: Drug: Pembrolizumab; Drug: Olaparib

INTERVENTIONS:
Drug: Pembrolizumab — pembrolizumab 200 mg every three weeks (Q3W)
  Other Names: KEYTRUDA
Drug: Olaparib — olaparib 300 mg twice daily (BID)
  Other Names: LYNPARZA

SUMMARY:
This trial is a multicenter, single-arm, phase 2 study of pembrolizumab in combination with olaparib in recurrent or metastatic cervical cancer patients who had disease progression during or after platinum-based chemotherapy.

DETAILED DESCRIPTION:
This trial is a multicenter, single-arm, phase 2 study of pembrolizumab in combination with olaparib in recurrent or metastatic cervical cancer patients who had disease progression during or after platinum-based chemotherapy.

This study is planned to enroll 28 patients eligible for participation from multiple study sites in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are at least 20 years of age on the day of signing informed consent with histologically confirmed, recurrent or metastatic cervical cancer (squamous cell carcinoma, adenocarcinoma or adenosquamous cell carcinoma)
2. Participants with confirmed disease progression during or after platinum-based chemotherapy 1 or intolerant to or ineligible for platinum-based chemotherapy or ineligible participants
3. Participants with measurable disease based on RECIST 1.1 at screening
4. Participant is able to provide a core or excisional biopsy of a tumor lesion for testing of PD-L1 status, etc
5. Participants with Eastern Cooperative Oncology Group (ECOG) PS of 0 to 1 upon the screening
6. Participants who may be expected to survive at least for 12 weeks after the first dose of study drug as determined by the principal investigator or a subinvestigator
7. Have adequate organ function

Exclusion Criteria:

1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
2. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to the enrollment.
3. Has received prior radiotherapy within 2 weeks prior to the enrollment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
4. Has received a live vaccine within 28 days prior to the enrollment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
5. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the enrollment.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the enrollment.
7. Has a second malignancy advanced or requiring treatment within the past 3 years.The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, in situ cancers (e.g. in situ breast carcinomas).
8. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to the enrollment.
9. Has severe hypersensitivity (≥Grade 3) to the study drug and/or any of its excipients.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and participants can be enrolled in the trial.
11. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a known history of Human Immunodeficiency Virus (HIV) infection.
14. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
15. Has a known history of active TB (Bacillus Tuberculosis).
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Participant has received colony-stimulating factors (eg, granulocyte colony stimulating factor [G-CSF], granulocyte macrophage colony-stimulating factor [GM-CSF] or recombinant erythropoietin) within 2 weeks prior to the enrollment.
18. Participant with clinically serious cardiovascular/cerebrovascular diseases including the following: cerebrovascular accident/stroke (less than 6 month prior to enrollment), myocardial infarction (less than 6 month prior to enrollment), unstable angina, congestive heart failure (the New York Heart Association (NYHA) Functional Classification Class 2 or severer), or serious arrhythmia. In addition, participants with history of bleeding tendency or recent major bleeding event in whom study drug administration carries higher risks as determined by the principal investigator will be excluded.
19. Participant who have acute or chronic disease with severe and/or clinical symptoms which may compromise the tolerance to this study or competence to consistently follow the study procedures as determined by the principal investigator
20. Participants with medical history of receiving all the PARP inhibitors
21. Participant is currently receiving either strong (eg, itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil) inhibitors of cytochrome P450 (CYP)3A4 that cannot be discontinued before the study drug initiation. The required washout period prior to starting olaparib is 2 weeks.
22. Participant is currently receiving either strong (eg, phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine, and St John's Wort) or moderate (eg. bosentan, efavirenz, modafinil) inducers of CYP3A4 that cannot be discontinued before the study drug initiation. The required washout period prior to starting olaparib is 5 weeks for phenobarbital and 3 weeks for other agents.
23. Participant is either unable to swallow orally administered medication or has a gastrointestinal disorder affecting absorption (eg, gastrectomy, partial bowel obstruction, malabsorption).
24. Participant has resting electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg, unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or participant has congenital long QT syndrome.
25. Has a major surgery history 4 weeks prior to the enrollment (e.g.: diagnostic biopsy is not regarded as the major surgery)
26. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
27. Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study, starting with the screening visit within 120 days after the last dose of trial treatment.
28. Participant, in the judgement of the investigator, is unlikely to comply with the study procedures, restrictions, and requirements of the study.
29. Participant has had an allogenic tissue/solid organ transplant

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 3 years
  Objective Response Rate (ORR) will be evaluated after pembrolizumab in combination with olaparib based on RECIST 1.1.

SECONDARY OUTCOMES:
Objective Response Rate on iRECIST | 3 years
  To assess ORR after administration of pembrolizumab in combination with olaparib based on iRECIST.
Duration of response | 3 years
  To assess duration of response (DOR) after administration of pembrolizumab in combination with olaparib based on RECIST 1.1 and iRECIST.
Durable response rate | 3 years
  To assess durable response rate (DRR) after administration of pembrolizumab in combination with olaparib based on RECIST 1.1 and iRECIST
Percentage of patients with response to administration of pembrolizumab in combination with olaparib for 6 months and longer | 3 years
  To assess the percentage of patients with response to administration of pembrolizumab in combination with olaparib for 6 months and longer based on RECIST 1.1 and iRECIST
PFS after administration of pembrolizumab in combination with olaparib | 3 years
  To assess progression-free survival (PFS) after administration of pembrolizumab in combination with olaparib based on RECIST 1.1 and iRECIST
Incidence of treatment-related adverse events after administration of pembrolizumab in combination with olaparib | 3 years
  To assess the number of participants with treatment-related adverse events after administration of pembrolizumab in combination with olaparib based on CTCAE v5.0
Objective Response Rate based on PD-L1 status | 3 years
  ORR will be evaluated after pembrolizumab in combination with olaparib stratified by PD-L1 status based on RECIST 1.1 and iRECIST.
Duration of response based on PD-L1 status | 3 years
  To assess DOR after administration of pembrolizumab in combination with olaparib stratified by PD-L1 status based on RECIST 1.1 and iRECIST.
Durable response rate based on PD-L1 status | 3 years
  To assess DRR after administration of pembrolizumab in combination with olaparib stratified by PD-L1 status based on RECIST 1.1 and iRECIST.
PFS based on PD-L1 status | 3 years
  To assess PFS after administration of pembrolizumab in combination with olaparib stratified by PD-L1 status based on RECIST 1.1 and iRECIST.

OTHER OUTCOMES:
Overall survival after administration of pembrolizumab in combination with olaparib based on RECIST 1.1 | 3 years
  To assess overall survival (OS) after administration of pembrolizumab in combination with olaparib based on RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Kosei Hasegawa, MD, PhD, Principal Investigator — Saitama Medical University International Medical Center
Locations (1):
- Saitama Medical Uiversity International Medical Center, Hidaka, Saitama, Japan

IPD SHARING:
Plan to Share IPD: No